CLINICAL TRIAL: NCT04130529
Title: Better Sleep in Psychiatric Care - Bipolar. A Randomized Naturalistic Study of a Psychological Group Treatment for Sleep Problems in Psychiatric Patients With Bipolar Disorder
Brief Title: Better Sleep in Psychiatric Care - Bipolar
Acronym: BSIP-Bipolar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Susanna Jernelöv, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/80-31/1
Record Dates: First submitted 2019-10-11; First posted 2019-10-17 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Sleep Problem; Bipolar Disorder
Keywords: Cognitive Behaviour Therapy; Psychological Intervention
MeSH Terms: conditions — Parasomnias; Bipolar Disorder | interventions — MD1

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjusted group CBT-i for Bipolar disorder (Experimental): The experimental group receives group-CBT-i adjusted for Bipolar disorder. This is a version of CBT for insomnia (CBT-i) developed during the pilot phase of this Project. Traditional CBT-i is adjusted for use in the population with Bipolar Disorder. This behavioral intervention adresses not only traditional aspects of insomnia, but also sleep phase problems and other aspects of sleep specifically relevant to the Bipolar population.
  Treatment is given as 8 weekly group sessions.
  Interventions: Behavioral: Adjusted group CBT-i for Bipolar disorder
- Sleep lectures (Active Comparator): The control group is offered a series of 3 lectures on sleep during the same time-period.
  Interventions: Other: Sleep lectures

INTERVENTIONS:
Behavioral: Adjusted group CBT-i for Bipolar disorder — CBT-i includes sleep scheduling/sleep compression, stimulus control, relaxation, cognitive interventions and sleep hygiene advice. In addition components targeting circadian rhythm problems and problems with very high or very low levels of activity are included.
  Arms: Adjusted group CBT-i for Bipolar disorder
Other: Sleep lectures — Lectures on the topic of sleep.
  Arms: Sleep lectures

SUMMARY:
Cognitive Behavioral Therapy (CBT) is treatment of choice for insomnia. Many patients in psychiatric care have sleep problems including insomnia, but are rarely given the choice to participate in CBT to improve their sleep. Patients with Bipolar disorder is a patient group with high levels of sleep difficulties. Sleep problems in this patient group can be both more general such as insomnia, but can also be related to the Bipolar disorder. Other research groups have studied the use of behaviorally sleep treatments in patients with Bipolar disorder, but more studies are needed. In a previous pilot study, the investigators of the current study developed a CBT protocol that would target sleep problems in this population. The basis was CBT for insomnia (CBT-i), but with more emphasis on achieving sleep promoting behaviors specific to Bipolar patients, for instance techniques that would also alleviate sleep phase problems, (e.g. the systematic use of light and darkness), and techniques to target more general sleep related problems (e.g. difficulties waking up in the morning), that are also common in patients with Bipolar disorder. This treatment was well tolerated and gave moderate effects on insomnia severity in the pilot study. In a naturalistic randomized controlled trial, the investigators now evaluate the effects of this psychological treatment on sleep and Bipolar symptoms in patients at the departments of Affective disorders, Northern Stockholm Psychiatry and Southwest Psychiatry, Stockholm, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient at the clinics involved in the project
* Experiencing sleep problems (subjective report)
* Being able to participate in a psychological intervention in group format

Exclusion Criteria:

* Night shift work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Changes from base-line to 8 weeks, 5 months and 14 months
  7-item, self-rated questionnaire measuring change in insomnia severity. Total score 0-28, higher score indicates more severe sleep problems.

SECONDARY OUTCOMES:
WHO Disability Assessment Schedule (WHODAS) | Changes from base-line to 8 weeks, 5 months and 14 months
  12-items self-rating questionnaire measuring disability. Total score (0-48), with higher score indicating more severe disability.
Affective Self Rating Scale (AS-18) | Changes from base-line to 8 weeks, 5 months and 14 months
  18-items self-report questionnaire measuring bipolar symptoms. Total score 0-72, subscale for depression (0-36), subscale for mania (0-36). Higher score indicates more severe symptoms.
Sleep habits and behaviors | Changes from base-line to 8 weeks, 5 months and 14 months
  Self-rating questionnaire regarding the use of sleep promoting behaviors. The questionnaire was constructed for the larger BSIP project and consists of two parts. The first part includes statements such as "Last week I got out of bed within 15 minutes of waking up" to be answered by number of days the last week this was true (i.e. from 0 to 7). The other part is to be answered on a 6-point Likert scale from "Not at all true" to "Entirely true", with 7 statements like "I get out of bed the same time every morning". No total score is obtained.
Daytime Insomnia Symptoms | Changes from base-line to 8 weeks, 5 months and 14 months
  7-item self-rating questionnaire regarding daytime symptoms commonly associated with sleep problems. Total score 0-70, with higher score indicating more severe daytime symptoms.
Actigraphy | Changes from base-line to post 8 weeks.
  An actigraph is placed on the participant's arm for one week. It measures participants' arm-movements. An algorithm can be used to estimate sleep from movement data.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Jernelöv, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Department of Affective Disorders, Northern Stockholm Psychiatry, Stockholm
  - Department of Affective Disorders, Stockholm Southwest Psychiatry, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan KA, Talavera DC, Harvey AG. Rise and shine: A treatment experiment testing a morning routine to decrease subjective sleep inertia in insomnia and bipolar disorder. Behav Res Ther. 2018 Dec;111:106-112. doi: 10.1016/j.brat.2018.10.009. Epub 2018 Oct 27. PMID 30399503
- [Background] Harvey AG, Soehner AM, Kaplan KA, Hein K, Lee J, Kanady J, Li D, Rabe-Hesketh S, Ketter TA, Neylan TC, Buysse DJ. Treating insomnia improves mood state, sleep, and functioning in bipolar disorder: a pilot randomized controlled trial. J Consult Clin Psychol. 2015 Jun;83(3):564-77. doi: 10.1037/a0038655. Epub 2015 Jan 26. PMID 25622197
- [Background] Kaplan KA, Harvey AG. Behavioral treatment of insomnia in bipolar disorder. Am J Psychiatry. 2013 Jul;170(7):716-20. doi: 10.1176/appi.ajp.2013.12050708. PMID 23820830